CLINICAL TRIAL: NCT01478620
Title: An Open-label, Non-randomized, Multicenter, Interventional Study to Investigate the Safety and Efficacy of Canephron® N in the Management of Uncomplicated Urinary Tract Infections (uUTI)
Brief Title: Safety and Efficacy of Canephron® N in the Management of Uncomplicated Urinary Tract Infections (uUTI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CanUTI2; 2011-000838-11 (EudraCT Number)
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

ARMS (1):
- Canephron® N (Experimental)
  Interventions: Drug: Canephron® N

INTERVENTIONS:
Drug: Canephron® N — 3x 2 coated tablets/day for 7 days p.o.

SUMMARY:
The objective of the study is to assess safety and impact of a non-antibiotic therapy approach with Canephron® N in the management strategy of uncomplicated lower urinary tract infections (UTIs).

DETAILED DESCRIPTION:
250 patients total 7-day treatment period with Canephron® N (2 tablets three times a day) and a follow-up period until Day 37. A total of three visits are planned on Day 0 (screening, start of study treatment), Day 7 (end of study treatment) and Day 37 (end of study visit).

Additional visits can be performed anytime between Day 1 and Day 37 if deemed necessary by the investigator. In case the patients experience consistent or worsening of symptoms they may be offered antibiotic therapy at the discretion of the investigator at any time. In this case Canephron® N intake will be stopped.

At least 50% of the patients, i.e. 125 subjects, should have received a 7-day treatment with Canephron® N. If less subjects are available recruitment of subjects will be continued until the required number of 125 subjects is reached.

Due to withdrawal of study in Russia total study population was reduced to 125 patients.

ELIGIBILITY:
Main Inclusion Criteria:

* Female outpatients aged 18-65 years (both inclusive).
* Patients suffering of symptoms of uncomplicated lower urinary infection at screening. Patients must have a total sum score of at least six for the symptoms dysuria, frequency and urgency.
* Development of symptoms within a maximum of 6 days before screening.
* Willing to refrain from consuming prohibited concomitant medications and products.
* Non-lactating female patients, who are surgically sterile (have had a documented bilateral oophorectomy and/or hysterectomy) or postmenopausal (cessation of menses for more than 1 year), or patients of childbearing potential with a negative pregnancy test at screening willing to use effective contraception methods (intrauterine device [IUD], hormonal contraceptives) during the study.

Main Exclusion Criteria:

* Any signs evoking complicated UTI, pyelonephritis and/or concomitant vulvo-vaginitis
* Any conditions that may lead to complicated infections (that is, renal diseases, urinary tract abnormalities or past urinary surgery, urine catheterization, etc).
* Chronic infection of the urinary tract requiring an intravenous pyelogram (IVP), ultrasound or cystoscopy.
* Current signs or symptoms of severe, progressive or uncontrolled life-threatening systemic disease i.e. renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease.
* Other acute infection (except UTI) requiring antibiotic treatment.
* Patients receiving treatment for presumed or proven urinary tract infection within 4 weeks prior to study entry.
* Antibiotic, immunosuppressive or immunostimulant (incl. vaccines) therapy within 4 weeks prior to study entry.
* Patients with known history of anatomical genitourinary (GU) anomalies or GU surgery within 6 months prior to study entry.
* Patients with known clinically significant abnormalities in screening physical examination, laboratory tests or vital signs.
* Peptic ulcers and hypersensitivity and/or idiosyncrasy to centaury herb, lovage root, rosemary leaves or one of the other ingredients of the investigational medicinal product.
* Rare hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency, galactose intolerance or lactase deficiency.
* Patients with a history of severe drug allergy or hypersensitivity.
* Known Human Immunodeficiency Virus (HIV)-seropositivity.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Ivanov, Principal Investigator — Kiev regional city hospital
Locations (1):
- Kiev Regional City Hospital, Kiev, Ukraine

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Canephron® N
Started | 125
Completed | 119
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Canephron® N
Number analyzed (Participants) | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 123
  >=65 years | 2
Sex/Gender, Customized [Number; unit: participants] — female participants
  participants | 125
Region of Enrollment [Number; unit: participants]
  Ukraine | 125
uncomplicated urinary tract infection symptom score [Mean (Standard Deviation); unit: score on a scale] — The severity of uUTI symptoms was assessed daily by the patient as well as by the investigator at each study visit. The following uUTI symptoms were rated on a 5-point scale: dysuria, frequency, urgency, acute development of incontinence or worsening of incontinence, nocturia, pain or discomfort in lower abdomen or pelvic areas and increased body temperature.
  The assessment of the symptoms ranged from 0 (absent or </= 37°C) to 4 (very severe or >/= 40°C).
  At baseline the total sum score (sum of subscales) of the symptoms dysuria, frequency and urgency had to be at least >/= 6.
  score on a scale | 7.3 (1.25)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Drug Reactions During 7-day Treatment of uUTI Symptoms With Canephron® N
Description: No study drug related adverse drug reactions were registered.
Time Frame: During active treatment period (day 1 until day 7)
Measure: Number; unit: Adverse Drug Reactions
Arm/Group | Canephron® N
Number analyzed (Participants) | 125
Adverse Drug Reactions | 0

2. Secondary Outcome: Incidence of Adverse Drug Reactions During the 7-day Treatment of uUTI Symptoms With Canephron® N in the Subgroup of Patients Who Take Canephron® N for at Least 7 Days
Time Frame: During active treatment period
Reporting Status: Not Posted

3. Secondary Outcome: Proportion of Patients With no Symptoms Worse Than Mild on Day 7 (i.e. Responders)
Time Frame: Day 7
Reporting Status: Not Posted

4. Secondary Outcome: Severity of uUTI Symptoms on Day 7
Time Frame: Day 7
Reporting Status: Not Posted

5. Secondary Outcome: Severity of uUTI Symptoms on Day 37
Time Frame: Day 37
Reporting Status: Not Posted

6. Secondary Outcome: Duration of uUTI Symptoms
Time Frame: During active treatment and follow up period (Day 0 - Day 37)
Reporting Status: Not Posted

7. Secondary Outcome: Proportion of Patients Who Require Antibiotic Treatment Until Day 7
Time Frame: During active treatment period
Reporting Status: Not Posted

8. Secondary Outcome: Proportion of Patients With Early Recurrence [Days] After Clearance of uUTI Symptoms
Time Frame: During active treatment and follow up period (Day 0 - Day 37)
Reporting Status: Not Posted

9. Secondary Outcome: Time to First Early Recurrence [Days] After Clearance of uUTI Symptoms
Time Frame: During active treatment and follow up period (Day 0 - Day 37)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Canephron® N
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 11/125
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Canephron® N (N=125)
Headache (Nervous system disorders) | 5 (9)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Heart rate irregular (Investigations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each Party acknowledges that it shall not publish any results of the trial,without the prior written authorization of the other Party. If SPONSOR (S.) requests INVESTIGATOR (I.)to publish any results obtained from the study, I. shall prepare and accomplish such publication at the expense of S. after review by S. and subject to written approval of the S. prior to publication. I. must be mentioned as co-author in any kind of publication resulting from such a request by S. to I. to publish.